CLINICAL TRIAL: NCT01353664
Title: An Open Label, Single-Arm Rollover Study for Subjects Who Participated In Other Romidepsin Protocols
Brief Title: A Rollover Study for Patients Who Participated in Other Romidepsin Protocols
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMI-ADVM-004; 2010-023040-32 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma; Cancer
Keywords: rollover protocol; romidepsin; Gloucester Pharmaceuticals; Celgene Corporation; continuing treatment
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin (Experimental): This study is an open-label, single-arm study. The study is divided into the Screening Period, Treatment Period, and Follow-up Period.
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — The participants will generally continue at the same dose, infusion time and frequency used for the last dose of romidepsin given in the preceding romidepsin study. If the participant entered this rollover study in the middle of a cycle, then the cycle number and cycle day will be carried over from the preceding romidepsin study.
  Other Names: Istodax®, ROMI

SUMMARY:
This study is intended to provide access to Romidepsin for participants who received Romidepsin in other trials sponsored by Gloucester Pharmaceuticals or Celgene Corporation and for participants whom the investigator feels may benefit from continuing treatment with Romidepsin.

DETAILED DESCRIPTION:
Participants must have previously participated in a Romidepsin study sponsored by Gloucester Pharmaceuticals or Celgene Corporation.

ELIGIBILITY:
Inclusion Criteria

1. Previously participated in and fulfilled the inclusion and exclusion criteria in one of the romidepsin clinical trials: ROMI-ADVM-001 (NCT01324310), ROMI-ADVM-002 (NCT01324323). Additional studies added at the discretion of the medical monitor of the study
2. Physician believes continued romidepsin treatment is of benefit to participant.
3. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
4. Able to adhere to the study visit schedule and other protocol requirements.
5. Negative urine or serum pregnancy test for females of child bearing potential; and
6. All females of child bearing potential must use an effective method of contraception (an intrauterine contraceptive device [IUCD] or double contraceptive method using condoms and a diaphragm plus spermicide) during the treatment period and for at least 1 month thereafter. Male participants should use contraception during the treatment period and for at least 3 months thereafter. Female participants should avoid the use of estrogen-containing contraceptives, since romidepsin may reduce the effectiveness of estrogen-containing contraceptives. An in vitro binding assay determined that romidepsin competes with β-estradiol for binding to estrogen receptors.

Exclusion Criteria

1. Concomitant use of drugs that may cause a significant prolongation of the corrected measurement of the time between the start of cardiac Q wave and the end of the T wave (QTc) .
2. Concomitant use of Cytochrome P 450 3A4 (CYP3A4) strong inhibitors within 1 week of trial medications.
3. Concomitant use of therapeutic warfarin due to a potential drug interaction. Use of a low dose of warfarin or another anticoagulant to maintain patency of venous access port and cannulas is permitted.
4. Prior chemotherapy or radiotherapy or any investigational agent after the last dose of romidepsin from the preceding romidepsin study.
5. Participants who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2012-09-05 (Actual); Study Completion 2012-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Takeshita, MD, Study Director — Celgene Corporation
Locations (3):
- United States (2):
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Sarah Cannon Research UK, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This rollover study was designed to give access to Romidepsin (Romi) for participants in and then discontinued from Romi studies ROMI-ADVM-001 (NCT01324310) and ROMI-ADVM-002 (NCT01324323) who in the opinion of the investigator could have benefited from ongoing therapy with Romi; those from GPI-06-0002 did not rollover as the study did not close.
Pre-assignment Details: Participants started at any point during a cycle which corresponded to their previous Romi study, but continued cycle numbering where it left off from their previous participation in a Romi study
Groups:
- ROMI 4: Participants received the same dose and frequency used for the last dose of romidepsin given in the preceding romidepsin study (either 8 mg/m^2 or 14 mg/m^2 on Days 1, 8 and 15 of a 28-day cycle), adjusted for any dose-limiting toxicities. For participants treated with the 4-hour infusion in their preceding romidepsin study, a change in the infusion time to 1-hour, at the dose/schedule of 10 mg/m^2 on Days 1, 8, and 15 every 28 days, was permitted upon consultation and agreement with the medical monitor.
Period: Overall Study
Arm/Group | ROMI 4
Started | 19 (Participants who received at least 1 dose of study drug.)
Completed | 0 (Completed = Number of participants who continued on Romidepsin treatment)
Not Completed | 19
Not completed — Other | 3
Not completed — Disease Progression | 16

BASELINE CHARACTERISTICS:
Arm/Group | ROMI 4
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (12.69)
Age, Customized [Number; unit: Participants]
  ≤ 65 | 10
  > 65 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black or African American | 1
  White | 15
  Other (unspecified) | 1
ECOG-Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a particpant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  Participants
    0 = Fully Active (Most Favorable Activity) | 9
    1 = Restricted activity but ambulatory | 10
    2 = Ambulatory; unable to carry out activities | 0
    3 = Limited Self-Care | 0
    4 = Completely Disabled | 0
Height [Mean (Standard Deviation); unit: Centimeters] — The total number for this baseline characteristic was 18; 1 participants' height was missing.
  Centimeters | 170.4 (11.02)
Weight [Mean (Standard Deviation); unit: Kilograms] — The number of participants with weight measured was 15; 3 were missing.
  Kilograms | 75.1 (20.06)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. Adverse events were assessed using National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4: On the following is the scale: Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe and Undesirable AE, Grade 4 = Life-threatening or Disabling AE, and Grade 5 = Death. Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention. A TEAE is defined as any AE occurring or worsening on or after the first dose of study drug and within 28 days after the last dose of study drug.
Time Frame: All AEs were recorded by the Investigator from the time the participant signed the informed consent to 28 days after the last dose of study drug; maximum drug exposure was 231 days
Population: Safety Population = Participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | ROMI 4
Number analyzed (Participants) | 19
Participants
  ≥ 1 Adverse Event (AE) | 18
  ≥ 1 AE related to study drug | 14
  ≥ 1 NCI CTCAE Grade 3 AE | 11
  ≥ 1 NCI CTCAE Grade 4-5 AE | 0
  ≥ 1 NCI CTCAE Grade 3 AE related to study drug | 6
  ≥ 1 NCI CTCAE Grade 4-5 AE related to study drug | 0
  ≥ 1 Serious Adverse Event (SAE) | 6
  ≥ 1 SAE related to study drug | 1
  ≥ 1 AE leading to discontinuation | 1
  ≥ 1 AE leading to stopping the study drug | 0
  ≥ 1 AE leading to dose reduction/interruption | 7
  ≥1 AE dose reduction related to study drug | 4

ADVERSE EVENTS:
Time Frame: All AEs were recorded by the Investigator from the time the participant signed the informed consent to 28 days after the last dose of study drug. Maximum time on study drug was 231 days
Arm/Group | ROMI 4
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ROMI 4 (N=19)
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Metastatic Carcinoma of the Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mental Status Changes (Psychiatric disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ROMI 4 (N=19)
Fatigue (General disorders) | 11
Asthenia (General disorders) | 4
Pyrexia (General disorders) | 4
Chills (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperlipidiaemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Ageusia (Nervous system disorders) | 1
Encephalopthy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Weight Decreased (Investigations) | 2
Electrocardiogram T Wave Inversion (Investigations) | 1
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Eye Swelling (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor that restricts the PIs rights to publish trial results after the trial is completed. Upon investigator submission of a publication to Celgene, Celgene will complete its review within 60 days after receipt of the publication. Upon Celgene's request, the publication shall be delayed up to 90 additional days to enable Celgene to secure intellectual property protection that would be affected by such proposed publication.